CLINICAL TRIAL: NCT04894643
Title: Preoperative, Proton- Radiotherapy Combined With Chemotherapy for Borderline Resectable Pancreatic Cancer
Acronym: PARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EBG MedAustron GmbH (Industry)
Collaborators: Landesklinkum Wiener Neustadt (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PARC-MA-062019
Record Dates: First submitted 2021-05-10; First posted 2021-05-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer; Proton Therapy
Keywords: Proton therapy combined with chemotherapy; Borderline Resectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Protons; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Capecitabine

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label, feasibility trial with gemcitabine and nab-paclitaxel, followed by concomitant proton therapy and capecitabine, followed by re-evaluation and surgery (when feasible) for patients with borderline resectable pancreatic cancer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative, proton- radiotherapy combined with chemotherapy (Other): Patients treated with three cycles of chemotherapy with Nab-PACLitaxel (Abraxane®) (125 mg/m² on day 1, 8, 15; powder for making a infusion solution) and Gemcitabine (1000 mg/m² on day 1, 8, 15; powder for making a infusion solution), followed by concomitant chemotherapy with capecitabine (1.660ml/m² on 5 days per week during the radiation therapy) and proton-therapy (with simultaneous integrated boost (SIB) 50.4 Gy Relative Biological Effectiveness (RBE) and 60.2 Gy (RBE) in 28 fractions of 1.8 Gy (RBE) and 2.15 Gy (RBE) 5 days per week), followed by re-evaluation and surgery
  Interventions: Radiation: Proton Ions; Drug: Nab-PACLitaxel; Drug: Gemcitabine; Drug: Capecitabine; Procedure: Surgical resection of the pancreas (when feasible)

INTERVENTIONS:
Radiation: Proton Ions — According to the radiation plan (between 50.4 and a maximum of 60.2 Gy) after Chemotherapy with Nab-PACLitaxel (Abraxane®) + Gemcitabine and concomitant to Capecitabine.
Drug: Nab-PACLitaxel — Chemotherapy will be delivered upfront for three cycles (week 2-4, week 6-8 and week 10-12) with combined Nab-PACLitaxel (Abraxane®) and Gemcitabine Therapy.
  It will be administered as intra venous infusion over 30 minutes.
  Other Names: Abraxane®
Drug: Gemcitabine — Chemotherapy will be delivered upfront for three cycles (week 2-4, week 6-8 and week 10-12) with combined Nab-PACLitaxel (Abraxane®) and Gemcitabine Therapy.
  Gemcitabine will also be administered as intra venous infusion over 30 minutes immediately after Nab-PACLitaxel.
Drug: Capecitabine — Concomitant to proton-radiotherapy (on the same days, within week 14-19)
Procedure: Surgical resection of the pancreas (when feasible) — Pre surgical re-evaluation will be performed at week 21 after enrollment. Patients fulfilling surgery-entry criteria, which consist of no distant metastasis, no massive ascites, no massive pleural effusion, no serious infection, no serious, unresolved chemoradiotherapy related, adverse events and adequate organ system function, will undergo surgery on week 22 (± 1 week). This should be performed via laparotomy.

SUMMARY:
This is an interventional, single arm, open-label, feasibility trial with gemcitabine and nab-paclitaxel, followed by concomitant proton therapy and capecitabine, followed by re-evaluation and surgery (when feasible) for patients with borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
This is an interventional, single arm, open label, feasibility trial of preoperative chemotherapy + concomitant chemo-proton therapy followed by surgery (when feasible) for patients with borderline resectable pancreatic cancer. Aim of this study is to test referral and enrollment procedures as well as technical feasibility. Proton therapy will be delivered in MedAustron, which is a stand alone facility. Pancreatic cancer patients are typically complex cases that require multidisciplinary care. Moreover delivery of high dose of proton therapy to large volumes including the upper abdomen lymphnodes and pancreatic neural plexus is technically challenging, therefore a feasibility study is deemed necessary. Following this study, a larger study will be performed aiming to confirm the ability of preoperative chemotherapy + concomitant chemo-proton therapy to improve resectability and ultimately outcome of borderline resectable pancreatic cancer without increase in toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis of pancreatic cancer
* Diagnosis of borderline resectable cancer according to the international consensus definition 2017.
* Negative staging for distant metastasis
* Blood test within the following limits absolute neutrophil count > 1,500 cells/mm³, platelet count > 100,000 cells/mm³, Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) < 2.5 times the upper limit of normal, total bilirubin < 2.5 times the upper limit of normal if patient had recent biliary stenting, total bilirubin < 1.5 times the upper limit of normal if no biliary stenting was done, serum creatinine within normal range (0.6-1.5 mg/dl) with a creatinine clearance > 30 ml/min (as estimated by Cockroft Gault equation)
* Age > 18 years
* Karnofsky index ≥ 70
* No tumor infiltration of stomach or duodenum
* The patient is informed of the diagnosis and is able to give informed consent (Ability of subject to understand character and individual consequences of the study protocol)
* Women of fertile age must have adequate conception prevention measures and must not breast feed
* Signed Informed Consent (must be available before study inclusion)

Exclusion Criteria:

* Non-exocrine tumors
* Major medical or psychiatric comorbidities that contraindicate radiation therapy, chemotherapy or surgery
* Presence of distant metastasis
* Pregnancy or unwilling to do adequate conception prevention
* Lactating and unwilling to discontinue lactation
* Men of childbearing potential not willing to use effective means of contraception
* Known allergic/hypersensitivity reaction to any of the components of study treatments
* Previous diagnosis of another neoplasm with worse prognosis as compared with the one in this study
* Metallic prosthesis or other condition that prevent an adequate imaging for target volume definition
* Loco-regional conditions that contraindicate radiotherapy e.g. active infections in the area
* Previous abdominal radiotherapy
* Prior systemic treatment for pancreatic cancer
* Hypersensitivity to PACLitaxel, albumin, gemcitabine or to any of the excipients of the chemotherapy
* Severe hepatic impairment
* Baseline Neutrophil Counts < 1.5 x 10^9/L
* Baseline Grade ≥ 2 sensory or motor neuropathy
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity - Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | from enrollment to six months after surgery
  Incidence of CTCAE version 5.0 Grade 4 non hematological toxicity from enrollment to six months after surgery
Perioperative Mortality and Complications | 90 days postoperatively
  Incidence of 90-days-perioperative mortality and incidence of Clavien Dindo Grade III complication rate during hospitalization

SECONDARY OUTCOMES:
Toxicity - CTCAE v5.0 | from enrollment to six months after surgery
  CTCAE V5.0 toxicity from enrollment to six month after surgery
Tumor recurrence | 260 weeks after therapy
  local and loco-regional (i.e. in-field) tumor recurrence
Progression free survival | 260 weeks after therapy
  loco-regional progression-free survival
Overall survival | 282 weeks
  Overall survival
Pathologic tumor response | 260 weeks
  Assessment of pathologic tumor response to pre-operative combined proton- chemotherapy (R0 margin and N0, degree of tumor cell necrosis in the resected tumor specimen)
Radiologic response | 263 weeks after proton therapy
  Assessment of radiologic response of pre-operative chemoradiotherapy. Response to preoperative treatment will be scored with the Japan Pancreas Society (JPS) classification which is a synthesis from the Evans and College of American Pathologists classification (Grade 1: poor or no response to Grade 4: complete response)
Quality of Life questionnaire: Functional Assessment of Cancer Therapy - Hepatobiliary (FACT-Hep) | 282 weeks
  Patient reported Quality of Life (for assessing disease-related symptoms and health-related quality of life). The higher the score the better the Quality of Life.
Quality of Life questionnaire: European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-30) | 282 weeks
  Questionnaire developed to assess the quality of life of cancer patients. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / quality of life (QoL) represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of Life questionnaire: Brief Pain Inventory | 282 weeks
  The Brief Pain Inventory (BPI) is a measurement tool for assessing clinical pain.The interference items were now presented with 0-10 scales, with 0=no interference and 10=interferes completely.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Fossati, M.D., Principal Investigator — EBG MedAustron GmbH; Friedrich Längle, Prim., Univ. Doz., M.D., Principal Investigator — LK Wiener Neustadt, Department of Surgery
Locations (2):
- Austria (2):
  - EBG MedAustron GmbH, Wiener Neustadt, Lower Austria
  - Department of Surgery, LK Wiener Neustadt, Wiener Neustadt